CLINICAL TRIAL: NCT03217227
Title: Evaluating Myocardial Ischemia in Chest Pain Using Cardiovascular Magnetic Resonance (CMR) Imaging Exercise Bike
Brief Title: Evaluating Myocardial Ischemia in Chest Pain Using Exercise CMR
Acronym: EMPIRE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Heart Centre Singapore (Other)
Responsible Party: Sponsor
Other Study IDs: 2017/2123
Record Dates: First submitted 2017-07-11; First posted 2017-07-14 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-04

CONDITIONS: Ischemic Heart Disease; Coronary Artery Disease; Cardiovascular Diseases; Myocardial Ischemia; Coronary Heart Disease; Microvascular Coronary Artery Disease
MeSH Terms: conditions — Myocardial Ischemia; Coronary Artery Disease; Cardiovascular Diseases; Coronary Disease | interventions — Cardiac Catheterization

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Approximately 30mL of blood in total will be drawn, where 25mL (equivalent to 5 teaspoons) of blood will be drawn before the exercise stress test and 5mL (equivalent to 1 teaspoon) of blood will be drawn after the exercise stress test.
  Blood samples will be collected from all participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy Volunteer: Healthy Volunteers will undergo the following study procedures:
  1. Cardiovascular Magnetic Resonance Imaging with Exercise Bike
  2. Blood Sampling
  3. Activity and Lifestyle Questionnaires
  4. Fat Mass Measurement
  Interventions: Other: Cardiovascular Magnetic Resonance Imaging with Exercise Bike
- Patients with Stable Angina: Patients will undergo the following study procedures:
  1. Cardiovascular Magnetic Resonance Imaging with Exercise Bike
  2. Blood Sampling
  3. Cardiac Catheterization
  4. Activity, Lifestyle and Medication Compliance Questionnaires
  5. Fat Mass Measurement
  6. Retinal Photography (Optional)
  7. I123 MIBG scan (Optional)
  Interventions: Other: Cardiovascular Magnetic Resonance Imaging with Exercise Bike; Procedure: Cardiac Catheterization; Other: Retinal Photography (Optional); Diagnostic Test: I123 MIBG Scintigraphy (Optional)

INTERVENTIONS:
Other: Cardiovascular Magnetic Resonance Imaging with Exercise Bike — A rest scan is performed and a gadolinium contrast may be administered during the scan (depending on the kidney function). After the rest scan is completed, images of the subject's heart during exercise via cycling in the supine position, will be scanned.
  Other Names: Bike MRI; CMR stress protocol
Procedure: Cardiac Catheterization — It is a procedure to diagnose and treat cardiovascular diseases by inserting a long and thin tube known as a catheter into the artery or vein in the neck, groin or arm and threaded through the blood vessels to the heart.
  A coronary angiogram is also performed during the procedure where an invisible contrast dye (only visible in the X-rays) is injected through the catheter and X-ray images scanned will show the flow of the dye through the heart arteries to determine any blockages in the arteries.
  In the case where there is severe narrowings, fractional flow reserve (FFR) may be performed to measure the pressure in the coronary arteries.
  If there is no significant narrowing lesions, the interventionist may perform additional flow resistance measurements of the small vessels to further investigate the cause of angina
  Other Names: Coronary Angiogram; Fractional Flow Resistance Measurement (FFR); Index of Microvascular Resistance Measurement (IMR); Coronary Pressure Measurement
  Groups: Patients with Stable Angina
Other: Retinal Photography (Optional) — The test studies the structure and function of the eye vessels. It involves using eye drops to dilate the pupils, allowing the retinal photographer to have a better view of the back of the eye.
  Groups: Patients with Stable Angina
Diagnostic Test: I123 MIBG Scintigraphy (Optional) — The test studies the cardiac sympathetic signalling that may help to identify patients with high risks of adverse events. The scan consists of 2 acquisitions of images 3-4 hours apart.
  For this study, only patients without clinically significant lesions (diagnosed via the cardiac catetherisation and have normal FFR results) will undergo this test.
  Other Names: Iodine-123-metaiodobenzylguanidine scintigraphy
  Groups: Patients with Stable Angina

SUMMARY:
Ischemic Heart Disease (IHD) is a condition of recurring chest pain or discomfort that occurs when a part of the heart is not receiving sufficient blood flow. It is a major public health concern internationally and in Singapore, the leading cause of death from cardiovascular disease. Cardiovascular magnetic resonance (CMR) has the ability to assess heart structures, scarring or lack of blood supply to the heart muscle with great accuracy and without any radiation involved. A CMR-compatible cycle ergometer can offer a safe and low cost stress equipment to assess heart function and motion abnormalities, and restrictions of the blood supply to the heart tissues due to partial or complete blockages of the blood vessels.

This study aims

1. to develop an exercise-CMR stress protocol by testing its feasibility and robustness in assessing changes in cardiac volumes and function due to physical exertion in healthy individuals and
2. to assess the accuracy of the multiparametric stress-CMR as a diagnostic tool for ischemic-causing coronary artery disease (CAD) with coronary fractional flow reserve (FFR) as a reference.
3. to measure the overall economic impact of ischaemic heart disease by estimating the direct and indirect medical costs for each participant. The current sample costs will be extrapolated to estimate the annual costs of treating and managing ischaemic heart disease in the local population.
4. to evaluate the effects of coronary microvascular dysfunction on coronary flow and regulation, physiological response and cardiac sympathetic signaling in patients with chest pain.

DETAILED DESCRIPTION:
Suspected ischemic heart disease (IHD) or coronary artery disease (CAD) is commonly diagnosed by stress testing where patients undergo exercise tests in order to make their hearts work hard and beat fast to require more blood and oxygen. Pharmacological-induced stress is employed in the case where the patient is unable to exercise. Since plaque-narrowed arteries cannot supply enough oxygen-rich blood to meet the heart's needs, the stress test can show signs and symptoms of IHD. Some of the symptoms include abnormal changes in the heart rate or blood pressure, shortness of breath, chest pain, or abnormal changes in the heart's rhythm and electrical activity.

As part of the stress tests, images of the heart are taken while the patient is exercising and while the patient is at rest. The imaging stress tests will show how well the blood flows in and out of the heart. An example would be a stress echocardiogram where an ultrasound is performed on the chest to produce video images of the heart to. IHD is detected through development of new regional wall motion abnormalities or worsening of preexisting regional wall motions. The patient will be required to exercise on a treadmill before lying on the examination bed for the ultrasound scan. This however, would require the patient to move from the treadmill to the bed, which would result in some time delay.

Another diagnostic test commonly used to diagnose IHD would be a nuclear scan known as myocardial perfusion imaging where a radioactive isotope acting as a tracer is injected into the bloodstream. During exercise, the tracer is monitored while it flows through the heart and lungs to allow detection for any blood-flow problems. However, this test would involve ionizing radiation due to the radioactive isotopic tracer used.

A detailed test to view blood flow through the heart, would be through a cardiac catheterization or an angiogram where a thin and flexible tube known as a catheter is threaded through an artery, usually in the leg, to the heart arteries. An invisible dye is injected through the catheter and special x-rays will be taken while the dye flows through the coronary arteries, allowing the doctor to study the blood flow through the heart and blood vessels. Due to the nature of the catheterization with the insertion of the tube, it makes the procedure invasive and hence involving risks although they are rare.

Cardiovascular magnetic resonance (CMR) is able to accurately and non-radiatively assess the heart structure, any scarring or lack of blood supply to the heart muscle. A CMR-compatible cycle ergometer offers a one-stop diagnostic test that is non-radiative and non-invasive. Hence, our investigators aim to develop a protocol that does not require any invasive procedure by assessing its accuracy and develop reference ranges in healthy individuals.

ELIGIBILITY:
Inclusion Criteria:

Healthy Volunteers:

* 21 years and above
* Normal physical examination
* No known significant medical history
* Able to give informed consent

Patients:

* 21 years and above
* Stable angina or angina-equivalent
* Has at least one of the following risk factors:

  1. Smoking
  2. Diabetes (fasting glucose level > 140 mg/dL)
  3. Hyperlipidemia (total cholesterol level > 250 mg/dL)
  4. Abnormal ECG
  5. Hypertension

Exclusion Criteria:

Healthy Volunteers:

* Contraindications to CMR implantable devices, cerebral aneurysm clips, cochlear implants
* Claustrophobia
* Women who are pregnant
* Inability to comply with study protocol
* Not able to exercise

Patients:

* Unstable cardiac conditions that are deemed by primary investigator to be unsuitable for this study
* Prior coronary revascularization or percutaneous coronary intervention
* Pulmonary disease
* Anemia
* Asthma
* Hyperthermia
* Hyperthyroidism
* Sympathomimetic toxicity
* Polycythemia
* Severely uncontrolled hypertension despite being on at least 3 anti-hypertensive medications

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The major source of recruitment for healthy volunteers will be from an existing database of healthy volunteers who have participated in the biobank program and have indicated interest in future studies. Other sources include co-workers of the department who volunteer and indicate on the Informed Consent Document that their participation was entirely voluntary and not coerced. Study Team members are ineligible.
  The major source of recruitment for patients with stable angina will be from the imaging and admission databases of the National Heart Centre Singapore. Patients are also referred by their attending healthcare professionals. The primary physicians of the patients identified will be notified and recruitment will only proceed if the primary physician is agreeable.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2017-05-01 (Actual); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
First occurrence of cardiovascular event | One year
  The outcomes are obtained via hospital records or phone follow-ups

CONTACTS AND LOCATIONS:
Overall Officials: Le Thu Thao, PhD, Principal Investigator — National Heart Research Institute Singapore
Locations (1):
- National Heart Centre Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Le TT, Ang BWY, Bryant JA, Chin CY, Yeo KK, Wong PEH, Ho KW, Tan JWC, Lee PT, Chin CWL, Cook SA. Multiparametric exercise stress cardiovascular magnetic resonance in the diagnosis of coronary artery disease: the EMPIRE trial. J Cardiovasc Magn Reson. 2021 Mar 4;23(1):17. doi: 10.1186/s12968-021-00705-8. PMID 33658056